CLINICAL TRIAL: NCT02178501
Title: The Effect of Omega-3 Polyunsaturated Acids Supplementation on Endothelial Function, Oxidative Stress, Platelet Aggregation, Blood Coagulation and Inflammation in Patients With Type 2 Diabetes and Cardiovascular Disease
Brief Title: Omega-3 Fatty Acids Supplementation and Atherothrombotic Biomarkers in Type 2 Diabetes and Cardiovascular Disease.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jagiellonian University (Other)
Collaborators: National Science Centre, Poland (Other Government)
Responsible Party: Principal Investigator, dr Grzegorz Gajos, prof.assoc., Jagiellonian University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 2011/03/B/NZ5/05767
Record Dates: First submitted 2014-04-12; First posted 2014-06-30 (Estimated); Last update posted 2016-11-29 (Estimated); Status verified 2016-11

CONDITIONS: Type 2 Diabetes; Cardiovascular Diseases
Keywords: OMEGA-3 PUFA; type 2 diabetes; cardiovascular diseases
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Cardiovascular Diseases | interventions — Docosahexaenoic Acids

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Omega-3 PUFA (Experimental): OMEGA-3 PUFA 2000 mg once daily (1000 mg EPA and 1000 mg DHA)
  Interventions: Dietary Supplement: Omega-3 PUFA
- Placebo (Placebo Comparator): Placebo once daily
  Interventions: Dietary Supplement: Omega-3 PUFA

INTERVENTIONS:
Dietary Supplement: Omega-3 PUFA — comparison of omega-3 PUFA supplementation 2000 mg once daily (1000 mg EPA and 1000 mg DHA) versus placebo

SUMMARY:
The major source of mortality and morbidity of diabetic patients is cardiovascular disease (CVD). Moreover, in CVD patients the presence of diabetes is associated with the increased risk of major adverse cardiac events as compared to patients without diabetes. The pathophysiology of macrovascular complications in T2D is not fully understood and involves: 1/ induction of oxidative stress, 2/ the formation of advanced glycation end products, 3/ activation of blood coagulation and platelet aggregation, 4/ increased inflammation, 5/ altered secretion of adipokines in obese subjects and 6/ endothelial dysfunction. All those mechanisms in T2D patients could potentially be a subject of new therapeutic interventions.

A therapy that continues to show promise in T2D patients with CVD is supplementation with omega-3 polyunsaturated fatty acids (PUFA). Clinical studies have indicated that omega-3 PUFA decrease the risk of major cardiovascular events, although the mechanism of action is not completely understood. Moreover, there were no trials exploring the mechanisms and outcomes of omega-3 treatment in T2D patients with CVD. Despite that fact, Polish Diabetes Association guidelines recommend the use of omega-3 PUFA in patients with diabetes in the prevention of macrovascular complications. Moreover, it is unclear whether the benefits of modifying the pathophysiological processes during supplementation with omega-3 PUFA occur only in patients with their deficiency or in all patients with type 2 diabetes.

Potential benefits of omega-3 PUFA in such patients are: 1/ decreased oxidative stress, 2/ decreased platelet aggregation and reduction of hypercoagulable state, 3/ anti-inflammatory effects, 4/ improvement in endothelial function. All those effects were explored previously with inconsistent findings. There is very limited information from clinical studies on the mechanisms and benefits of omega-3 PUFA in T2D patients with CVD.

The objective of the current study is to evaluate the effects of omega-3 PUFA administered on top of optimal therapy of atherosclerotic vascular disease and T2D on endothelial function, platelet aggregation and thrombotic, inflammatory and oxidative stress biomarkers.

DETAILED DESCRIPTION:
The study will provide insight into:

1. The influence of the baseline level of omega-3 PUFA in patients with type 2 diabetes mellitus (T2D) and CVD on endothelial function, platelet aggregation and thrombotic, inflammatory, oxidative stress biomarkers.
2. The potential to improve the endothelial function, reduce the oxidative stress and to decrease the atherothrombotic and inflammatory biomarkers with the supplementation with a moderate dose of omega-3 PUFA
3. The mechanisms of the clinically observed effects of omega-3 PUFA in T2D patients with CVD.

SCIENTIFIC BACKGROUND The incidence of diabetes is growing in the world and the number of patients already exceeded 360 million and by 2030 this will rise to 552 million. The major source of mortality and morbidity of diabetic patients is cardiovascular disease (CVD). On average, it is estimated that people with type 2 diabetes (T2D) will die 5-10 years before people without T2D, mostly due to CVD. The treatment of CVD accounts for a large part of the huge healthcare costs attributable to T2D (10-12% of European health care expenditure). Despite significant improvements in the treatment of CVD with antiplatelet agents, statin, angiotensin converting enzyme inhibitors (ACEI) and newer antidiabetic drugs the mortality of diabetic patients with CVD is continuously significantly higher than in people without T2D. This pattern of elevated cardiovascular risk in diabetes has been attributed to several possible mediating factors, including the development of more extensive, multi-vessel coronary artery disease, the presence of impaired myocardial systolic contractility, diffuse small vessel endothelial dysfunction and the presence of a hypercoagulable or pro-thrombotic state attributable to diabetes.

The increased cardiovascular risk in T2D patients is generated by the metabolic disturbances related to diabetes (both hyperglycaemia and hypoglycaemia) and that includes:

* irreversible glycation of intra- and extracellular proteins leading to changes in gene expression and induction of oxidative stress leading to endothelial dysfunction,
* activation of protein kinase C resulting in activation of blood coagulation,
* increase in the levels of various pro-atherothrombotic and inflammatory biomarkers e.g. markers of platelet activation, thrombin generation, endothelin, von Willebrand factor, adhesion molecules (eg.VCAM-1, vascular endothelial cell adhesion molecule), growth factors (VEGF), factor VII, CRP, IL-6 (interleukin-6). Moreover it was recently described that hyperglycemia in T2D leads to nonenzymatic glycation of fibrinogen. Glycated fibrinogen leads to denser fibrin clots that are stiffer and more resistant to fibrinolysis, thus leading to an increased thrombotic burden,
* altered secretion of adipokines by adipose tissue in obese subjects with T2D. It was demonstrated that greater adiposity e.g. down-regulates secretion of adiponectin, an adipokine with anti-inflammatory and insulin-sensitizing properties.

All those pro-atherothrombotic mechanisms in T2D patients could potentially be a subject of new developments in the treatment, especially in patients with CVD. A therapy that continues to show great promise in this indication is supplementation with omega-3 polyunsaturated fatty acids (PUFA) although the underlying mechanism of their beneficial action is not precisely known. Numerous prospective and retrospective trials have shown that omega-3 PUFA supplementation decreases the risk of major cardiovascular events, such as myocardial infarction, sudden cardiac death, coronary heart disease, atrial fibrillation, and most recently, death in patients with heart failure. However, none of those trials was performed in T2D patients with CVD who are at the highest risk of events and where benefits could have considerable clinical importance. Moreover to our knowledge, there are very few randomized, double-blind, placebo-controlled clinical trials exploring the mechanisms of omega-3 treatment in T2D patients with documented cardiovascular disease. Despite that fact, Polish Diabetes Association guidelines recommend the use of omega-3 PUFA in patients with diabetes in the prevention of macrovascular complications. Moreover, it is unclear whether the benefits of modifying the pathophysiological processes during supplementation with omega-3 PUFA occur only in patients with their deficiency or in all patients with type 2 diabetes.

Although there are several potential benefits considering therapy with omega-3 PUFA in T2D patients with atherosclerotic vascular disease, some of those effects require a detailed appraisal in a clinical study. They are:

1. Platelet activation and resistance to antiplatelet agents. Platelet dysfunction in diabetes mellitus is related to several mechanisms - including metabolic derangements, oxidative stress, and endothelial dysfunction. They lead to high platelet reactivity which has been associated with atherothrombotic complications in patients with T2DM. Therefore antiplatelet therapy is one of the cornerstones of secondary prevention of atherothrombotic events in patients with T2DM.

   Recent evidence suggests that the clinical efficacy of both aspirin and clopidogrel is compromised in subjects in diabetes by mechanisms that are not entirely clear. This is one of the reasons why diabetic patients continue to have a higher risk of adverse cardiovascular events compared with that in non-diabetic patients.

   The antiplatelet effect of n-3 PUFA has been explored with inconsistent findings. Recently, the investigators have demonstrated that the addition of n-3 PUFA to the combination of aspirin and clopidogrel significantly potentiates platelet response to clopidogrel after percutaneous coronary intervention (PCI).

   So far, there are no studies evaluating the effects of n-3 PUFA on platelet reactivity and response to antiplatelet agents in patients with T2D and CVD.
2. Coagulation and fibrinolysis. In patients with T2D there is a general increase in plasma levels of procoagulant factors accompanied by a decreased fibrinolytic capacity.

   The mechanisms for these alterations are complex, with insulin resistance and hyperglycaemia being clear culprits. The net result of the above changes is an increased tendency to clot formation, with the fibrin network displaying a compact structure and resistance to fibrinolysis. Moreover, increased fibrinogen levels observed in diabetes correlate with the degree of hyperglycemia and with fibrinogen glycation affecting fibrin polymerization and factor XIII-mediated crosslinking. Of note, impaired metabolic control and marked fluctuations in plasma glucose levels have been shown to be related to hypofibrinolysis associated with the formation of dense fibrin clots. The differences in fibrin clot structure and its susceptibility to lysis found to occur in type 2 diabetes may contribute to the increase in CVD risk in diabetic patients.

   A number of measures can reduce the hypercoagulable environment in diabetes including glycaemic control, with avoidance of hypoglycaemia and improvement in insulin sensitivity. Of the pharmacological agents used in patients with T2D and CVD, metformin, aspirin, statins and angiotensin converting enzyme inhibitors have a favourable effect on the coagulation system and all have been shown to reduce cardiovascular events in diabetes.

   Although it is unclear whether n-3 PUFA has clinically relevant effects on insulin resistance in humans, they may affect coagulation system directly via several mechanisms. It has been shown that in apparently healthy subjects, omega-3 PUFA can increase or decrease plasma fibrinogen and clotting factors, in particular factor VII activity, factor VIII and von Willebrand factor concentrations. There are studies indicating that fish oil supplementation may reduce thrombin generation. Conversely, other studies failed to demonstrate significant changes in circulating markers of thrombosis following administration of omega-3 PUFA. Of note, these studies have been conducted in patients without diabetes, so the knowledge on the effects of omega-3 in T2D patients with CVD treated on optimal pharmacotherapy (including drugs affecting the coagulation) is limited.

   Regarding the effects of omega-3 PUFAs on fibrinolytic activity the findings are controversial. In a single study performed 20 years ago intake of omega-3 PUFAs has been associated with increased plasma plasminogen activator inhibitor (PAI-1) activity in non-insulin-dependent diabetes mellitus patients. Interestingly, in a recent study, PAI-1 concentration and activity increased more following high omega-3 PUFAs beverage compared with low omega-3 PUFAs beverage in men with metabolic syndrome. It was also demonstrated that with respect to fibrinolytic measurements, acute and chronic intake of fish oil may show opposite effects, although the underlying mechanistic basis for this is not understood. Further research is needed on this potentially adverse effect on the coagulation in patients with glycometabolic disorders.
3. Endothelial dysfunction and oxidative stress A large body of evidence links endothelial dysfunction to human diabetes mellitus. Endothelial dysfunction in T2D contributes to the pathogenesis and clinical expression of atherosclerosis by promoting inflammation, thrombosis, arterial stiffness, and impaired regulation of arterial tone and flow.

   Increased oxidative stress in the vasculature is an important mechanism of endothelial dysfunction and insulin resistance in diabetes mellitus. For example, circulating markers of oxidative stress, including F2 isoprostanes and antibodies against oxidized low density lipoprotein, are increased in humans with T2D.

   In recent years, growing evidence links the intake of omega-3 PUFA with an improvement in endothelial function. The mechanisms by which omega-3 PUFAs might influence endothelial function are likely to be multiple and complex. They could include the suppression of thromboxane A2 or cyclic endoperoxides, a reduced production of cytokines, the augmented endothelial synthesis of nitric oxide, an improvement of vascular smooth muscle cell sensitivity to nitric oxide, and a reduced expression of endothelial adhesion molecules. The reduction of oxidative stress with omega-3 PUFA in patients with T2D may be an important factor responsible for the improvement of endothelial function. However, there is not enough data on the improvement of endothelial function and the reduction of oxidative stress in patients with T2D and established CVD.
4. Inflammation Chronic inflammation may participate in the pathogenesis of insulin resistance, type 2 diabetes, and cardiovascular disease and may be a common denominator that links obesity to these disease states. A variety of circulating proinflammatory cytokines and acute-phase reactants are increased in obesity, type 2 diabetes, and cardiovascular disease. Moreover, chronic low-grade inflammation occurring in the adipose tissue of obese individuals is linked to increased insulin resistance and leads to disturbances in the adipokines secretion.

Although there are divergent data whether omega-3 PUFA reduce inflammation they may modulate adipokine secretion from adipose tissue. It was demonstrated that they increase plasma adiponectin levels, which could be a potential mechanism by which EPA and DHA improve insulin sensitivity. They also induce leptin and visfatin secretion and reduce the expression of several proinflammatory cytokines from the adipose tissue, including tumor necrosis factor TNFα, IL-6, monocyte chemotactic protein MCP-1, and PAI-1. However, there are no clinical studies whether omega-3 PUFA supplementation can modulate adipose tissue inflammation in T2D patients with CVD.

ELIGIBILITY:
Inclusion Criteria:

* min. 50 years old at screening
* type 2 of diabetes diagnosed for at least 6 months (regardless of the mode of hypoglycemic therapy)
* HbA1c ≥ 6,5%
* concomitant coronary artery disease (with significant, reversible or irreversible myocardial perfusion defect, providing existing ischemia or history of myocardial infarction) or cerebrovascular or peripheral vascular disease (documented with angiography)

Exclusion Criteria:

* pregnancy
* type 1 diabetes or poorly controlled T2D (HbA1c > 9.0%)
* acute myocardial infarction within less than 3 months
* percutaneous coronary intervention, coronary artery bypass grafting, percutaneous transluminal angioplasty or vascular surgery within less than 1 month
* acute infection
* hypertriglyceridemia requiring treatment with omega-3 PUFA
* active bleeding or any known coagulation or bleeding disorders
* concomitant chronic anticoagulant therapy
* platelet count < 100x109/L
* serum creatinine > 177 μmol/L (2 mg/dL)
* liver injury (alanine transaminase level > 1.5 times above the upper limit of the reference range)
* chronic use of nonsteroidal anti-inflammatory drugs other than aspirin
* daily intake of dietary supplements containing omega-3 PUFA within the past month
* known sensitivity or allergy to fish or omega-3 fatty acid supplements
* history of inflammatory disease or vasculitis or corticosteroid therapy
* active substance abuse
* history of malignancy (unless disease free for >10 years, or non-melanoma skin carcinoma)
* projected life-expectancy <12 months due to comorbid condition
* any abnormal laboratory value or physical finding that according to the investigator may interfere with the interpretation of the study results, be indicative of an underlying disease state, or compromise the safety of a potential subject

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2013-01; Primary Completion 2015-12 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in biomarkers of oxidative stress at 3 months | From baseline to 3 months
  8-iso-prostaglandin F2α, oxidized LDL;
Change from Baseline in coagulation status at 3 months | From baseline to 3 months
  1. Platelet aggregation (induced by 5 and 20 μmol/L of adenosine diphosphate (ADP) and by 0.5 mmol/L of arachidonic acid; light transmittance aggregometry)
  2. Thrombin generation (prothrombin 1.2 fragments, endogenous thrombin potential)
  3. Platelet-fibrin clot strength measurements (thromboelastography)
  4. Fibrin clot properties (permeability and lysis)
Change from Baseline in endothelial function status 3 months | From baseline to 3 months
  1. Flow mediated vasodilation in brachial artery (FMD)
  2. Asymmetric Dimethylarginine (ADMA), ICAM-1, VCAM-1, von Willebrand factor

SECONDARY OUTCOMES:
Change from Baseline in fatty acids metabolism at 3 months | From baseline to 3 months
  1. Serum Phospholipid Fatty Acids
  2. total cholesterol, triglycerides, HDL-cholesterol, LDL-cholesterol
  3. adiponectin, leptin
Change from Baseline in glycometabolic control at 3 months | From baseline to 3 months
  1. Fasting glucose, HbA1c 2. Insulin, C-peptide 2. Homeostasis model assessment HOMA-IR

OTHER OUTCOMES:
Safety Measures | at 3 months
  1. Occurrence of any type of ischemic or bleeding complications
  2. Liver enzymes changes

CONTACTS AND LOCATIONS:
Overall Officials: Grzegorz Gajos, prof.assoc., Principal Investigator — Department of Coronary Disease, Institute of Cardiology, Jagiellonian University Medical College
Locations (2):
- Poland (2):
  - Samodzielny Publiczny Szpital Kliniczny nr 7 Śląskiego Uniwersytetu Medycznego w Katowicach Górnośląskie Centrum Medyczne im. prof. Leszka Gieca, Katowice
  - Krakowski Szpital Specjalistyczny im. Jana Pawła II, Krakow

REFERENCES:
- [Derived] Poreba M, Mostowik M, Siniarski A, Golebiowska-Wiatrak R, Malinowski KP, Haberka M, Konduracka E, Nessler J, Undas A, Gajos G. Treatment with high-dose n-3 PUFAs has no effect on platelet function, coagulation, metabolic status or inflammation in patients with atherosclerosis and type 2 diabetes. Cardiovasc Diabetol. 2017 Apr 14;16(1):50. doi: 10.1186/s12933-017-0523-9. PMID 28410617